CLINICAL TRIAL: NCT01706042
Title: Over-night Metabolic Effects of Legumes
Brief Title: Effects of Legumes on Glucose Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Anti-Diabetic Food Centre (Other)
Responsible Party: Principal Investigator, Anne Nilsson, assistant lector, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 668/2008
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Dietary Prevention

ARMS (2):
- white bread (Placebo Comparator): White bread (based on 35 g available carbohydrates)
  Interventions: Other: white bread
- Legume meal (Active Comparator): Legumes are consumed as a late evening meal(based on 35 g available carbohydrates)
  Interventions: Other: legume meal

INTERVENTIONS:
Other: legume meal
  Arms: Legume meal
Other: white bread
  Arms: white bread

SUMMARY:
Dietary prevention strategies are increasingly recognized as essential to combat the current epidemic of obesity and related metabolic disorders. The purpose of the present study was to evaluate the potential effects of legumes in relation to cardiometabolic risk markers and appetite regulating hormones.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 20-35 years
* With normal BMI and
* No known metabolic- or gastro intestinal disease

Exclusion Criteria:

* BMI > 25,
* Known metabolic disorder or
* Gastrointestinal problems or disease

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
blood glucose | 11 hours
  A portion of legumes or bread was consumed as a late evening meal, blood glucose was measured the next morning at breakfast.

SECONDARY OUTCOMES:
satiety | 11 hours
  legumes or bread was consumed as a late evening meal, satiety hormones (PYY, oxyntomodulin)and appetite sensations were determined at a following breakfast.

OTHER OUTCOMES:
inflammatory markers | 11 hours
  legumes or bread was consumed as a late evening meal, inflammatory markers (IL-6, IL-8)was determined at a following breakfast.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Nutrition and Food Chemistry, Lund University, Lund, Sweden

REFERENCES:
- [Background] Sievenpiper JL, Kendall CW, Esfahani A, Wong JM, Carleton AJ, Jiang HY, Bazinet RP, Vidgen E, Jenkins DJ. Effect of non-oil-seed pulses on glycaemic control: a systematic review and meta-analysis of randomised controlled experimental trials in people with and without diabetes. Diabetologia. 2009 Aug;52(8):1479-95. doi: 10.1007/s00125-009-1395-7. Epub 2009 Jun 13. PMID 19526214
- [Background] Papanikolaou Y, Fulgoni VL 3rd. Bean consumption is associated with greater nutrient intake, reduced systolic blood pressure, lower body weight, and a smaller waist circumference in adults: results from the National Health and Nutrition Examination Survey 1999-2002. J Am Coll Nutr. 2008 Oct;27(5):569-76. doi: 10.1080/07315724.2008.10719740. PMID 18845707
- [Derived] Nilsson A, Johansson E, Ekstrom L, Bjorck I. Effects of a brown beans evening meal on metabolic risk markers and appetite regulating hormones at a subsequent standardized breakfast: a randomized cross-over study. PLoS One. 2013;8(4):e59985. doi: 10.1371/journal.pone.0059985. Epub 2013 Apr 5. PMID 23577078